CLINICAL TRIAL: NCT06602999
Title: Addressing the Nutritional Needs of Cancer Survivors With Nutrition Insecurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24806; NCI-2024-07163 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); U54CA280811 (NIH)
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
Keywords: Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (Instacart voucher, nutrition navigation) (Experimental): Participation receive a booklet on nutrition and physical activity for cancer survivors and 1 Instacart grocery delivery voucher to use over 4 weeks on study. Participation also receive nutrition navigation phone calls for assistance with following nutrition guidelines and ordering groceries on Instacart every week for 4 weeks.
  Interventions: Other: Nutritional Intervention; Other: Instacart Voucher; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Nutritional Intervention — Receive a booklet on nutrition and physical activity for cancer survivors
Other: Instacart Voucher — Receive Instacart grocery delivery voucher
  Other Names: Nutritional Intervention
Behavioral: Telephone-Based Intervention — Receive nutrition navigation phone calls

SUMMARY:
This clinical trial studies whether the use of a grocery delivery service (Instacart) and nutrition navigation improves food insecurity in cancer survivors. The American Cancer Society recommends a normal body mass index, regular physical activity, and a healthy diet for cancer patients. Following these guidelines may help prevent deaths among cancer patients, but few cancer patients follow them. One reason for not following the guidelines could be due to the lack of consistent access to sufficient quantities of affordable, nutritious food for an active, healthy life (food insecurity). Instacart provides users access to foods that fall under the nutrition plan for cancer survivors that can be purchased and delivered to the user's home from many different grocery stores. Nutrition navigation provides support to cancer survivors via weekly check ins to help with following nutrition guidelines and assist with ordering groceries on the Instacart platform. Using a grocery delivery service, such as Instacart, and nutrition navigation may help improve food insecurity in cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the intervention's feasibility and acceptability.

SECONDARY OBJECTIVES:

I. To estimate the effect of the intervention on adherence to American Cancer society nutrition guidelines.

II. To estimate the effect of the intervention on self-reported food insecurity.

III. To evaluate the feasibility of patient navigation calls. IV. To evaluate the feasibility of Instacart vouchers.

EXPLORATORY OBJECTIVE:

I. To evaluate the feasibility of the intervention through an end-of-study semi-structured interview.

OUTLINE:

Patients receive a booklet on nutrition and physical activity for cancer survivors and 1 Instacart grocery delivery voucher to use over 4 weeks on study. Patients also receive nutrition navigation phone calls for assistance with following nutrition guidelines and ordering groceries on Instacart once a week (QW) for 4 weeks.

After completion of study intervention, patients are followed up at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of a malignant cancer (except non-melanoma skin cancer).
* Not on active treatment at the time of screening and not expected to receive active anticancer therapy (e.g., surgery, radiation, chemotherapy, immunotherapy, targeted therapies) during the study period. Hormonal therapies are allowed for patients with breast or prostate cancer
* At least 6 weeks since a major surgery and fully recovered.
* Have access to the internet and able to send and receive text messages.
* Able to speak/read English.
* Based on the United States Department of Agriculture (USDA) United States (U.S.) Household Food Security Survey, identify as experiencing food insecurity and/or belong to a population that the National Institutes of Health (NIH) has identified as being at risk for health disparities:

  * Identify as a racial or ethnic minoritized group, as defined by the NIH (American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Pacific Islander, Latino or Hispanic)
  * Identify with a sexual or gender minoritized group.
  * Annual household income < 200% of the federal poverty definition and/or education < bachelor's degree.
  * Live in a rural and/or a persistent poverty area (based on zip code).

Exclusion Criteria:

* Contraindication to any study-related procedure or assessment.
* Planned major surgery or cancer-directed therapy during the study period.
* Living outside of the US or Canada during screening and/or the study period (outside the geographic areas that Instacart covers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Median score on the Feasibility of Intervention Measure (FIM) score | 4 weeks
  The FIM is a four-item measure of implementation that assesses participants perceived appropriateness of the intervention. Each item response falls on a scale of 1 (Completely disagree) to 5 (Completely agree). A scaled score is calculated by averaging responses. Scale values range from 1 to 5. The intervention will be determined acceptable if the overall median score is >= 4. The median and (interquartile range (IQR) of the FIM score.
Median score on the Acceptability of Intervention Measure (AIM) score | 4 weeks
  The AIM is a four-item measure of implementation that assesses participants perceived acceptability of the intervention. Each item response falls on a scale of 1 (Completely disagree) to 5 (Completely agree). A scaled score is calculated by averaging responses. Scale values range from 1 to 5. The intervention will be determined acceptable if the overall median score is >= 4. The median and (IQR) of the AIM score.
Appropriateness of intervention measure (IAM) score | 4 weeks
  The IAM is a four-item measure of implementation that assesses participants perceived appropriateness of the intervention. Each item response falls on a scale of 1 (Completely disagree) to 5 (Completely agree). A scaled score is calculated by averaging responses. Scale values range from 1 to 5. The intervention will be determined acceptable if the overall median score is >= 4. The median and (IQR) of the AIM score.

SECONDARY OUTCOMES:
Change in intake of fruit and vegetables, whole grains, sugar sweetened beverages, red meat, and processed meat | Up to 4 weeks
  Will describe intake of fruit and vegetables, fiber, whole grains, added sugars, dairy, calcium, red meat, and processed meat from the dietary screeners at enrollment and end of study, as well as change in intake between time points, using medians (IQR). Will examine changes in dietary intakes and adherence to the American Cancer Society nutrition guidelines pre- to post-intervention using paired t-tests. Will use mean (95% CI) and median (IQR) to describe intakes at each time point and change over time.
Mean change in participant reported United States Department of Agriculture Food Insecurity score | Up to 4 weeks
  The United States Department of Agriculture Food Insecurity Questionnaire consists of 6 items that address various aspect of food security. Responses of "often" or "sometimes" and "yes" are coded as affirmative. Responses of "almost every month" and "some months but not every month" are coded as affirmative. The sum of affirmative responses to the six questions in the module is the household's raw score on the scale. Food security status is assigned as follows: Raw score 0-1 = High or marginal food security (raw score 1 may be considered marginal food security, but a large proportion of households that would be measured as having marginal food security using the household or adult scale will have raw score zero on the six-item scale), Raw score 2-4=Low food security, Raw score 5-6=Very low food security. The mean change in score over time will be reported.
Proportion of participants who completed navigation calls | Up to 4 weeks
  The proportion of participants who completed navigation calls will be reported.
Proportion of participants using Instacart vouchers | Up to 4 weeks
  The proportion of participants who utilized the Instacart vouchers during the course of the study will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Sorbarikor Piawah, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Zuckerberg San Francisco General, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets will be shared with research collaborators
Supporting Information: Study Protocol, SAP

DOCUMENTS (1):
  • Informed Consent Form (2025-03-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT06602999/ICF_000.pdf